CLINICAL TRIAL: NCT03338179
Title: Evaluation of Metamemory in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: LAPSCO, Psychology University, Blaise Pascal University, Clermont-Ferrand. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-360; 2010-A00857-32 (Other: 2010-A00857-32)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia; Aging
Keywords: Metamemory; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult Patients (Experimental): Schizophrenia patients aged between 18 and 45 years old
  Interventions: Behavioral: Judgement of learning evaluation
- Aged Patients (Experimental): Schizophrenia patients aged 59.5 years and above
  Interventions: Behavioral: Judgement of learning evaluation
- Adult Controls (Active Comparator): Controls aged between 18 and 45 years old
  Interventions: Behavioral: Judgement of learning evaluation
- Aged Controls (Active Comparator): Controls aged 59.5 years and above
  Interventions: Behavioral: Judgement of learning evaluation

INTERVENTIONS:
Behavioral: Judgement of learning evaluation — The hardware consists of two lists of 30 pairs of French words, each pair of words being composed of a word index and a target word (names of concrete objects). Among the 60 word pairs, 30 are strongly associated items (or easy items, the other 30 being weakly associated or difficult items.

SUMMARY:
The purpose of this study is to determine the respective roles of aging and schizophrenia in the regulation of metamemory using a generation strategy. 4 groups will be necessary to comparison:

Adult patients (18-45 years) Adult controls (18-45 years) Aged patients (≥ 59.5 years) Aged controls (≥ 59.5 years)

The effects of age and the disease could lead to interaction in regulating metamemory. The effect of age would be aggravated by the disease.

DETAILED DESCRIPTION:
Metamemory measurement

* Objective: Measurement of monitoring and control capabilities, and relations between these two abilities when learning of word pairs.
* Description: The hardware consists of two lists of 30 pairs of French words, each pair of words being composed of a word index and a target word (names of concrete objects). Among the 60 word pairs, 30 are strongly associated items (or easy items, the other 30 being weakly associated or difficult items.

In front of a computer screen, each participant is subjected to a learning test in which 30 pairs of words appear one by one on the screen. Participants have the option to control the time of presentation of each pair of words. After a retention time of 4 minutes of information devoted to nonverbal distractive task, follows an evaluation phase of deferred judgments of learning (JOL time), where for each pair of words studied, the word index is presented without the target word. Participants must then assess a learning judgment for each pair of words, that is to say they have to estimate, on a 5-point scale, their ability to remember later the target word in the presentation the index word. This JOL assessment phase is immediately followed by cued recall test.

For the second learning test (30 other word pair), the steps are identical. Prior to this second learning, generating instruction of a pair of words to learn is proposed: a word index is presented to the participants who have to generate a pair with a target word. Participants are trained on 5 pairs of words.

ELIGIBILITY:
Inclusion Criteria:

* For both:
* Age: between 18 and 45 years for adults, and 59.55 and above for older,

For patients :

* DSM-5 criteria of schizophrenia
* Adult patients (<45 years) will be matched to elderly patients (> 59.55 years) gender and educational level,
* Patients followed as outpatients,
* Age of onset of the disease less than 40 years,
* Patients whose disease has stabilized: no changes psychotropic treatment for at least 1 month
* Not more of a benzodiazepine,
* Patients on protection of justice or not,

For controls :

* - Matched for sex to patient
* Age-matched (+/- 3 years) to patient
* Matched for educational level (+/- 2 years) to patients

Exclusion Criteria:

* -For patients :
* Any other comorbid psychiatric diagnosis of Axis I DSM-5 (particularly depression, addiction excluding tobacco, dementia)
* Patients with impaired vision or hearing preventing the realization of the tests.
* Long-term Anticholinergic treatment.
* Patients with less 5 years of school

For controls:

* Any psychiatric diagnosis according to DSM-5, including addictions (excluding tobacco)
* Head injuries, brain injuries or diseases,
* vision or hearing problems preventing the realization of the tests.
* Current or past addiction to all toxic substances except tobacco.
* Long-term Anticholinergic treatment.
* Related to the first degree diagnosed with a psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2016-05-23 (Actual)

PRIMARY OUTCOMES:
difference of judgement of learning using a 5 point scale (0%, 25%, 50%, 75%, 100%) using a generation strategy. | at day 1
  the 4 groups of participants formed by the case-control study in two age strata value their judgments of learning for each pair of words using a 5 point scale (0%, 25%, 50%, 75%, 100%) with the generation strategy.

SECONDARY OUTCOMES:
Difference of judgement of learning using a 5 point scale (0%, 25%, 50%, 75%, 100%) between generation and reading strategies | at day 1
  the 4 groups of participants formed by the case-control study in two age strata, value their judgments of learning for each pair of words using a 5 point scale (0%, 25%, 50%, 75%, 100%) in a generation strategy and in a reading strategy.
Difference of number of recalled word using a generation strategy | at day 1
  the 4 groups of participants formed by the case-control study in two age strata recalled the word they learn using a generation strategy.
Difference of number of recalled word between generation and reading strategies | at day 1
  the 4 groups of participants formed by the case-control study in two age strata recalled the word they learn using a generation strategy and a reading strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle JALENQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France